CLINICAL TRIAL: NCT04783922
Title: An Update on Intracerebral Hemorrhage - A Cohort Study
Brief Title: An Update on Intracerebral Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shifa Clinical Research Center (Other)
Collaborators: Shifa International Hospital (Other); Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Junaid Akram, Dr. Muhammad Junaid Akram, Shifa Clinical Research Center
Other Study IDs: IRB-Approval- Submitted
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Intracerebral Hemorrhage; Stroke; Hematoma
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Hematoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Benign Hematoma: Patients (having novel image markers or clinical features) suggestive of a benign hematoma relatively , that is having relatively good prognostic outcome and less likely to expand.
- Malignant Hematoma: Patients (having novel image markers or clinical features) suggestive of a malignant hematoma relatively, that is more likely to expand and have poor prognostic outcome.

SUMMARY:
The intracerebral hemorrhage study is a multicenter , combination of prospective and retrospective observational cohort study led by Dr. Muhammad Junaid Akram, PhD scholar at Chongqing Medical University. Prof Dr. Qi Li will be the senior consultant for the study. The study will be focusing on natural history, epidemiological , radiological, rehabilitative and clinical aspects as well as the effect of various treatments on the hemorrhagic patients.

The study related data of the patients diagnosed with intracerebral hemorrhage will be collected in prospective and retrospective ways. The prognostic data for the patients will be assembled and collected via using different outcome measures at different points of time.

DETAILED DESCRIPTION:
The study will be used to address the several key issues related to intracerebral hemorrhage. The demographics, scores based upon disease severity , mRS, GCS, NIHSS scores will be recorded at baseline and in the prospective and retrospective ways. The data obtained from the registered patients will be used for future use , critical review by expert neurologists, neurorehabilitative experts for further use and review.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years Patients willing to participate via signing a consent form' Patients diagnosed with CT-Confirmed spontaneous intracerebral hemorrhage (ICH) Patients willing to participate in the follow up assessment

Exclusion Criteria:

* Not willing to participate Secondary ICH to hemorrhagic infarction or tumor bleeding etc. Traumatic ICH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprising of the participants willing to participate in the study with an age greater than 18 years from Pakistan.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
hematoma volume growth at 24 hours | 24 hours
  To assess early hematoma volume growth at 24 hours

SECONDARY OUTCOMES:
Functional outcome at 3 months assessed by modified Rankin Scale | 3 months
  Assess functional outcome at 3 months by using mRS
Early neurological deterioration assessed by NIHSS score at 24 hours | 24 hours
  To assess early neurological deterioration by using NIHSS score at 24 hours
Early neurological deterioration assessed by NIHSS score at 48 hours | 48 hours
  To assess early neurological deterioration by using NIHSS score at 48 hours
Early neurological deterioration assessed by NIHSS score at 72 hours | 72 hours
  To assess early neurological deterioration by using NIHSS score at 72 hours
Perihematomal edema volume measurement at 24 hours | 24 hours
  To measure the perihematomal edema volume growth at 24 hours
Perihematomal edema volume measurement at 48 hours | 48 hours
  To measure the perihematomal edema volume growth at 48 hours
Perihematomal edema volume measurement at 72 hours | 72 hours
  To measure the perihematomal edema volume growth at 72 hours
Intraventricular hemorrhage growth | 24 hours
  To assess the presence of IVH at 24 hours
Major thrombotic events | 2 weeks
  To assess the thrombotic events 2 weeks after admission

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Junaid Akram, DPT, MS-NMPT, Principal Investigator — Chongqing Medical University, Chongqing / Shifa Tameer e Millat University, Islamabad
Locations (1):
- Shifa Tameer e Millat University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet